CLINICAL TRIAL: NCT06957639
Title: Investigation of the Effects of Different Physiotherapy Approaches Applied to Patients With Chronic Non-Specific Neck Pain on Pain Level, Grip Strength and Manual Dexterity: A Randomized Controlled Trial
Brief Title: Physiotherapy in Chronic Neck Pain
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Kevser Gürsan, Principal Investigator, Uşak University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 585-585-07
Record Dates: First submitted 2025-04-26; First posted 2025-05-04 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Neck Pain
Keywords: neck pain; physiotherapy; manual dexterity; grip strenght
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: parallel single-blind randomized study
Who Masked: Outcomes Assessor
Masking Description: This study has a single-blind randomized controlled design. The applications will be applied directly to the participants by the researchers, but the person conducting the evaluations will be unaware (blind) of which participant is in which intervention group. The evaluator performing the measurements will not know the group assignments of the participants, thus minimizing the risk of bias in the measurement and evaluation processes.
  For this purpose, group information will be kept confidential during data collection and only the time of measurement and the participant ID code will be reported to the evaluator.
  Group identities will also be represented by codes during the data analysis phase, and group identities will be revealed after the analysis is completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Other): Group 1: Standard physiotherapy intervention and home exercises
  Interventions: Other: Standard physiotherapy intervention and home exercises
- Group 2 (Experimental): Group 2: Trigger point therapy and home exercises
  Interventions: Other: Trigger point therapy and home exercises
- Group 3 (Experimental): Group 3: Kinesiology Taping therapy and home exercises
  Interventions: Other: Kinesiology Taping therapy and home exercises
- Group 4 (Experimental): Group 4: Cervical - Scapular Mobilization and home exercises:
  Interventions: Other: Cervical - Scapular Mobilization and home exercises

INTERVENTIONS:
Other: Standard physiotherapy intervention and home exercises — Various physical agents such as electrotherapy, hotpack (warm compress) and ultrasound therapy will be used within the standard physiotherapy intervention. These approaches are effective methods to reduce pain, relax muscles and accelerate healing. Home exercises are daily neck exercises recommended by a specialist physiotherapist.
  Arms: Group 1
Other: Trigger point therapy and home exercises — Trigger point therapy is a common method used in patients with myofascial pain syndrome. This method involves manually releasing trigger points. Approaches such as pressure applications and stretching techniques are used. Muscle functions are improved by loosening painful muscle knots. Muscle flexibility and endurance are increased with home exercises.
  Arms: Group 2
Other: Kinesiology Taping therapy and home exercises — Kinesiology taping is an elastic band technique used for pain management and muscle activity support. It accelerates healing by increasing blood circulation. It supports and protects the muscles in the neck and shoulder area.
  It provides supportive stabilization without restricting joint movements. It facilitates movement by reducing pain. It targets muscle strengthening and mobilization with home exercises
  Arms: Group 3
Other: Cervical - Scapular Mobilization and home exercises — Cervical and scapular mobilization includes manual therapy techniques aimed at increasing the range of motion of the joints in the spine and shoulder area. Mobilization is applied to the cervical spine and shoulder joints. Relaxation is provided in the muscles around the shoulder and neck. Cervical and scapular stability is improved. Postural disorders are corrected and range of motion is increased. Sustainability of mobilization is ensured with home exercises.
  Arms: Group 4

SUMMARY:
In this randomized controlled experimental study design, it was aimed to examine whether different treatment approaches frequently applied in physical therapy clinics have an effect on pain, hand grip strength and hand skills by applying them to individuals with CNNP. For this purpose, the following hypotheses were created.

H1: Standard physiotherapy intervention and home exercises have an effect on reducing the pain intensity of individuals with CNNP H2: Standard physiotherapy intervention and home exercises have an effect on increasing the hand grip strength of individuals with CNNP.

H3: Standard physiotherapy intervention and home exercises have an effect on increasing the hand skills of individuals with CNNP.

H4: Trigger point therapy and home exercises have an effect on reducing the pain intensity of individuals with CNNP.

H5: Trigger point therapy and home exercises have an effect on increasing the hand grip strength of individuals with CNNP.

H6: Trigger point therapy and home exercises have an effect on increasing the hand skills of individuals with CNNP.

H7: Kinesiology Taping treatment and home exercises have an effect on reducing the pain intensity of individuals with CNNP.

H8: Kinesiology Taping treatment and home exercises have an effect on increasing the hand grip strength of individuals with CNNP.

H9: Kinesiology Taping treatment and home exercises have an effect on increasing the manual skills of individuals with CNNP.

H10: Cervical - Scapular Mobilization and home exercises have an effect on reducing the pain intensity of individuals with CNNP.

H11: Cervical - Scapular Mobilization and home exercises have an effect on increasing the hand grip strength of individuals with CNNP.

H12: Cervical - Scapular Mobilization and home exercises have an effect on increasing the manual skills of individuals with CNNP.

4 different groups will be created in this study. These are Group 1: Standard physiotherapy intervention and home exercises Group 2: Trigger point therapy and home exercises Group 3: Kinesiology Taping therapy and home exercises Group 4: Cervical - Scapular Mobilization and home exercises

DETAILED DESCRIPTION:
Neck pain is one of the musculoskeletal disorders with a high prevalence in the adult population. Its prevalence in the world varies between 16.7% and 75.1% and is generally more common in women than in men. Neck pain is a public health problem that should be considered in terms of individual health and general well-being as well as health expenditures. As a result of ignoring neck pain, neck pain becomes chronic. Neck pain, which significantly affects the quality of life of individuals with chronic neck pain (CNP), causes restrictions in movement and decreases in upper extremity functions. In particular, the functions of the hand, which are indicators of upper extremity functions frequently used in daily life activities, are the functions of the hand. Studies have found that individuals with chronic neck pain have decreased grip strength and psychomotor skills compared to healthy individuals. Based on this, various treatment methods have been applied to individuals with CNP in many similar studies in the literature to reduce the level of pain, prevent disability, increase performance in daily life activities and increase joint range of motion. There is no study that examines whether the various physical therapy methods frequently applied in this clinic have an effect on the grip strength and manual dexterity of individuals with CNNP by applying them together comparatively. In this context, four different groups will be formed for the research. The first group will receive standard physiotherapy intervention, the second group will receive trigger point therapy for the neck region, the third group will receive kinesiology taping, and the fourth group will receive cervical and scapular mobilization treatment methods. Individuals in all four groups will be advised to do daily home exercise programs and told to apply them. The applications will be applied four times a week for four weeks, for a total of 16 sessions. Then, before and after the application, neck pain levels of individuals with CNNP, fine hand skills evaluation, and grip strength measurements will be made. Thus, it will be found out whether these different treatment approaches will reduce the pain intensity of individuals with CNNP, whether grip strength, which is an important indicator of upper extremity performance, is increased, and whether fine hand skills will be improved. The purpose of this study; It will be determined whether different physiotherapy approaches applied to individuals with chronic nonspecific neck pain have an effect on the individuals' pain level, grip strength and manual skills. The results will reveal how different physiotherapy interventions can play a role in pain management and improving upper extremity performance in individuals with CNNP. Similar studies conducted today will be examined with the results we obtain and various solution suggestions will be presented.

ELIGIBILITY:
Inclusion Criteria:

* Being 18-64 years old,
* Having neck pain for 3 months or more,
* being literate, being a volunteer

Exclusion Criteria:

* having musculoskeletal injuries in the neck-shoulder area,
* having neurological or orthopedic problems,
* having cancer, having musculoskeletal malformations,
* having had head and neck surgery,
* having received physical therapy due to neck pain in the last 6 months
* not accepting to participate in the study,
* being pregnant,
* individuals with hearing and visual impairments

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2025-07-25 (Estimated); Study Completion 2025-07-25 (Estimated)

PRIMARY OUTCOMES:
Pain assessment | Four weeks
  Pain assessment will be made with Visual Analog Scale (VAS). VAS was developed by Price et al. in 1983 for the assessment of subjective pain and is a reliable and easy-to-apply scale that has been accepted in the world literature. VAS is a scale with two different names on the vertical or horizontal line, 10 cm long (0=I have no pain - I am very comfortable and 10=The most unbearable pain).

SECONDARY OUTCOMES:
Grip Strength Assessment | Four weeks
  Grip strength assessment will be done with Jamar hand dinanometer. Measurements will be made 3 times with the Hand Dynamometer and the average will be taken. Hand Dynamometer is accepted as the gold standard for measuring grip strength. Measurement will be made for both hands (right and left).
Fine motor skills assessment | Four weeks
  Fine manual dexterity assessment will be done with the Nine-Hole Peg Test. NHPT consists of a 9-hole platform and 9 rods. The platform will be placed directly in front of the individuals and the rods will be adjusted so that the holes are on the dominant hand side of the individuals and the holes are on the non-dominant hand side. After the test rules are explained to the individuals, they will be given the opportunity to practice before the application. Individuals will be asked to insert the rods into the board as quickly as possible. Test results will be recorded by measuring the time from the moment the individuals touch the first rod until the last rod is inserted into the platform with a stopwatch. Then, they will be asked to remove the 9 rods one by one with the same hand and the removal time will be recorded. The test will be applied to the non-dominant hand using the same method; this time, the platform will be rotated in front of the non-dominant hand.

CONTACTS AND LOCATIONS:
Overall Officials: Kevser Gursan, Dr., Principal Investigator — Uşak University
Locations (1):
- Yozgat Bozok University Health Application and Research Center, Yozgat, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
In order to protect participant confidentiality and comply with the confidentiality commitment approved by the ethics committee, no sharing of individual-level data is planned. In addition, the ethics committee decision that approved the study covers data use with limited access only. Therefore, it may not be possible to share IPD data publicly.